CLINICAL TRIAL: NCT05258513
Title: The Effects of Oral Supplementation With Geranylgeraniol (GG) Sourced From Annatto on Sexual Health in Males and Females
Brief Title: The Effects of Geranylgeraniol (GG) Sourced From Annatto on Sexual Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122102
Record Dates: First submitted 2022-02-04; First posted 2022-02-28 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Sexual Health; Libido
Keywords: Sexual Health; Libido; Body Composition; Strength; Vitality; Hormones

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel, randomized, placebo controlled, dose-escalation trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): From weeks 1-4, participants will consume 150mg daily of a visually identical placebo. For weeks 5-8, the dose will be escalated as participants will consume 300mg daily of placebo supplementation.
  Interventions: Dietary Supplement: Placebo Supplementation
- Geranylgeraniol Treatment (Experimental): From weeks 1-4, participants will consume 150mg daily of a Geranylgeraniol (GG). For weeks 5-8, the dose will be escalated as participants will consume 300mg daily of GG.
  Interventions: Dietary Supplement: GG sourced from Annatto

INTERVENTIONS:
Dietary Supplement: Placebo Supplementation — 8 weeks of placebo supplementation
  Arms: Placebo
Dietary Supplement: GG sourced from Annatto — 8-weeks of Geranylgeraniol supplementation
  Arms: Geranylgeraniol Treatment

SUMMARY:
The purpose of this study will be to examine the effectiveness of Geranylgeraniol supplementation on sexual health function in males and females following an 8-week dose escalation intervention. The study will be carried out in a randomized, double-blind, placebo-controlled, parallel manner. Participants will be stratified into quartiles based on their scores on the Derogatis Interview for Sexual Functioning during screening and prior to baseline testing. Participants from each quartile will be randomly divided by into treatment or placebo conditions.

Following randomization, participants will be baseline assessed on their sexual health function using a variety of questionnaires, body composition using a whole body Dual Energy X-Ray Absorptiometry scan, blood chemistry panel, and grip strength using a hand-held dynamometer. Following baseline testing, participants will undergo 8 weeks of supplementation of their respective supplement condition. Participants will be instructed to consume two servings a day (150mg total per day) from weeks 1-4. Subject will return to the study site after 4 weeks to reassess the above-mentioned parameters. Participants will then undergo a dose escalation and be instructed to consume two servings a day (300mg total per day) from week 5-8. Sexual health questionnaires and assessments of body composition, blood chemistry, and grip strength will be conducted following the week 8 to conclude the study.

DETAILED DESCRIPTION:
The purpose of this study will be to examine the effectiveness of Geranylgeraniol supplementation on sexual health function in males and females following an 8-week dose escalation intervention. The study will be carried out in a randomized, double-blind, placebo-controlled, parallel manner. Participants will be stratified into quartiles based on their scores on the Derogatis Interview for Sexual Functioning during screening and prior to baseline testing. Participants from each quartile will be randomly divided by into treatment or placebo conditions.

Following randomization, participants will be baseline assessed on their sexual health function using a variety of questionnaires, body composition using a whole body Dual Energy X-Ray Absorptiometry scan, blood chemistry panel, and grip strength using a hand-held dynamometer. Following baseline testing, participants will undergo 8 weeks of supplementation of their respective supplement condition. Participants will be instructed to consume two servings a day (150mg total per day) from weeks 1-4. Subject will return to the study site after 4 weeks to reassess the above-mentioned parameters. Participants will then undergo a dose escalation and be instructed to consume two servings a day (300mg total per day) from week 5-8. Sexual health questionnaires and assessments of body composition, blood chemistry, and grip strength will be conducted following the week 8 to conclude the study.

Participants will be assessed for the following variables on Week 0, 4, and 8:

Primary Variables:

Subjective measures related to sexual health by administering the following questionnaire in both Males and Females

* Derogatis interview for sexual functioning self report (DISF-SR)

Subjective measures to Male specific questionnaires:

* Aging Male Symptoms (AMS)
* Erectile Dysfunction Inventory for Treatment Satisfaction (EDITS)
* Erection Hardness Satisfaction (EHS)
* Index of Erectile Function (IIEF-5)
* Androgen Deficiency in Aging Male (ADAM) in those >40 years old

Subjective measures to Females specific questionnaires:

* Hot flashes and night sweats
* Female Sexual Function Index

Secondary variables:

* Bone density, lean mass, and body fat percentage via Dual Energy X-Ray Absorptiometry (DEXA)
* Hand grip strength assessed via handheld dynamometer
* Bioavailable and total testosterone, estradiol, progesterone, Dihydrotestosterone (DHT), and Sex Hormone Binding Globulin (SHBG) in blood serum

Subjective measures related to well-being via the following questionnaires:

* Quality of life (SF-36)
* Perceived stress scale 10 (PSS-10)
* Sleep quality index
* Multidimensional fatigue index
* International physical activity questionnaire (IPAQ)

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 30-49 years old
* Males scoring 27-36 on the Aging Males Symptoms scale
* Willing to sign the Informed Consent
* English literate

Exclusion Criteria:

* Cardiovascular, neurological, metabolic, or endocrine disease
* Drink heavily (>7 and >14 drinks per week for women and men, respectively)
* Smoke
* Renal, hematological, or hepatic disorder
* Psychiatric disorder, depression
* Peptic ulcer
* Any malignancy
* Thrombosis
* Undergone surgery that affects digestion and absorption
* Hypo- or hypertensive
* Undergoing hormone replacement therapy
* Using hormone boosting supplements (herbal or synthetic)
* Using drugs that are anti-diabetic, anti-platelet, anti-coagulant, beta blockers, or used to treat ED
* Pregnant or trying to conceive, currently breastfeeding, or have breastfeed within the prior 3 months
* Have participated in a clinical trial within the past 6 months

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2022-02-06 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in Overall Sexual Function | Week 0, 4 and 8
  Assessed by administering the Derogatis Interview for Sexual Functioning (DISF-SR) for subjective measurement. Values range from 0 to 8 with higher scores demonstrating a better outcome.
Changes in Aging Male Symptoms | Week 0, 4, and 8
  Assessed by administering the Aging Male Symptoms scale to males for subjective measurement. Values range from 1 to 5 with lower scores demonstrating a better outcome.
Changes in Androgen Deficiency in Aging Males Scale | Week 0, 4, and 8
  Assessed by administering the Androgen Deficiency in Aging Males scale to males for subjective measurement. Values range from 1 to 5 with higher scores demonstrating a better outcome.
Changes in Satisfaction to Treatment | Week 4 and 8
  Assessed by administering the Erectile Dysfunction Interview for Treatment Satisfaction (EDITS) to males for subjective measurement. Values range from 0 to 4 with lower scores demonstrating a better outcome.
Changes in Erection Hardness | Week 0, 4 and 8
  Assessed by administering the Erection Hardness Score (EHS) to males for subjective measurement. Values range from 0 to 4 with higher scores demonstrating a better outcome.
Changes in Erectile Function | Week 0, 4 and 8
  Assessed by administering the International Index of Erectile Function (IIEF) to males for subjective measurement. Values range from 0 to 5 with higher scores demonstrating a better outcome.
Changes in Female Sexual Function | Week 0, 4 and 8
  Assessed by administering the Female Sexual Function Index to females for subjective measurement. Values range from 0 to 5 with higher scores demonstrating a better outcome.
Changes in Hot Flashes | Week 0, 4 and 8
  Assessed by administering the Hot Flashes and Night Sweats questionnaire to females for subjective measurement. Values range from 0 to 10 with lower scores demonstrating a better outcome.
Changes in Night Sweats | Week 0, 4 and 8
  Assessed by administering the Hot Flashes and Night Sweats questionnaire to females for subjective measurement. Values range from 0 to 10 with lower scores demonstrating a better outcome.

SECONDARY OUTCOMES:
Testosterone | Week 0, 4, and 8
  Experimental outcome examining bioavailable and total testosterone in fasted whole blood samples
Estradiol | Week 0, 4, and 8
  Experimental outcome examining bioavailable and total estradiol in fasted whole blood samples
Progesterone | Week 0, 4, and 8
  Experimental outcome examining bioavailable and total progesterone in fasted whole blood samples
Sex Hormone Binding Globulin (SHBG) | Week 0, 4, and 8
  Experimental outcome examining total SHBG in fasted whole blood samples
Changes in Dihydrotestosterone (DHT) | Week 0, 4, and 8
  Experimental outcome examining total DHT in fasted whole blood samples
Changes in White Blood Cell count | Week 0, 4, and 8
  Experimental outcome examining total White Blood Cell count via fasted whole blood samples
Changes in Red Blood Cell count | Week 0, 4, and 8
  Experimental outcome examining total Red Blood Cell count via fasted whole blood samples
Changes in Hemoglobin levels | Week 0, 4, and 8
  Experimental outcome examining total Hemoglobin via fasted whole blood samples
Changes in Hematocrit levels | Week 0, 4, and 8
  Experimental outcome examining total Hematocrit via fasted whole blood samples
Changes in Mean Corpuscular Volume | Week 0, 4, and 8
  Experimental outcome examining total Mean Corpuscular Volume via fasted whole blood samples
Changes in Mean Corpuscular Hemoglobin | Week 0, 4, and 8
  Experimental outcome examining total Mean Corpuscular Hemoglobin via fasted whole blood samples
Changes in Mean Corpuscular Hemoglobin Concentration | Week 0, 4, and 8
  Experimental outcome examining total Mean Corpuscular Hemoglobin Concentration via fasted whole blood samples
Changes in Red Cell Distribution Width | Week 0, 4, and 8
  Experimental outcome examining total Red Cell Distribution Width via fasted whole blood samples
Changes in Platelet Count | Week 0, 4, and 8
  Experimental outcome examining total Platelet count via fasted whole blood samples
Changes in Mean Platelet Volume | Week 0, 4, and 8
  Experimental outcome examining total Mean Platelet volume via fasted whole blood samples
Changes in Granulocyte levels | Week 0, 4, and 8
  Experimental outcome examining percentage of Granulocytes via fasted whole blood samples
Changes in Lymphocytes levels | Week 0, 4, and 8
  Experimental outcome examining percentage of Lymphocytes via fasted whole blood samples
Changes in Monocyte levels | Week 0, 4, and 8
  Experimental outcome examining percentage of Monocytes via fasted whole blood samples
Changes in Eosinophil levels | Week 0, 4, and 8
  Experimental outcome examining percentage of Eosinophil via fasted whole blood samples
Changes in Basophil levels | Week 0, 4, and 8
  Experimental outcome examining percentage of Basophil via fasted whole blood samples
Changes in Granulocyte count | Week 0, 4, and 8
  Experimental outcome examining total Granulocyte via fasted whole blood samples
Changes in Lymphocytes count | Week 0, 4, and 8
  Experimental outcome examining total Lymphocytes via fasted whole blood samples
Changes in Monocyte count | Week 0, 4, and 8
  Experimental outcome examining total Monocytes via fasted whole blood samples
Changes in Eosinophil count | Week 0, 4, and 8
  Experimental outcome examining total Eosinophil via fasted whole blood samples
Changes in Basophil count | Week 0, 4, and 8
  Experimental outcome examining total Basophil via fasted whole blood samples
Changes in Glucose levels | Week 0, 4, and 8
  Experimental outcome examining total Glucose via fasted whole blood samples
Changes in Blood Urea Nitrogen levels | Week 0, 4, and 8
  Experimental outcome examining total Blood Urea Nitrogen via fasted whole blood samples
Changes in Serum Creatinine levels | Week 0, 4, and 8
  Experimental outcome examining total Serum Creatinine via fasted whole blood samples
Changes in Sodium levels | Week 0, 4, and 8
  Experimental outcome examining total Sodium via fasted whole blood samples
Changes in Potassium levels | Week 0, 4, and 8
  Experimental outcome examining total Potassium via fasted whole blood samples
Changes in Chloride levels | Week 0, 4, and 8
  Experimental outcome examining total Chloride via fasted whole blood samples
Changes in Carbon Dioxide levels | Week 0, 4, and 8
  Experimental outcome examining total Carbon Dioxide via fasted whole blood samples
Changes in Calcium levels | Week 0, 4, and 8
  Experimental outcome examining total Calcium via fasted whole blood samples
Changes in Total Protein levels | Week 0, 4, and 8
  Experimental outcome examining total Protein via fasted whole blood samples
Changes in Albumin levels | Week 0, 4, and 8
  Experimental outcome examining total Albumin via fasted whole blood samples
Changes in Globulin levels | Week 0, 4, and 8
  Experimental outcome examining total Globulin via fasted whole blood samples
Changes in Total Bilirubin levels | Week 0, 4, and 8
  Experimental outcome examining total Bilirubin via fasted whole blood samples
Changes in Alkaline Phosphatase levels | Week 0, 4, and 8
  Experimental outcome examining total Alkaline Phosphatase via fasted whole blood samples
Changes in Alanine Transaminase levels | Week 0, 4, and 8
  Experimental outcome examining total Alanine Transaminase via fasted whole blood samples
Changes in Aspartate Aminotransferase levels | Week 0, 4, and 8
  Experimental outcome examining total Aspartate Aminotransferase via fasted whole blood samples
Changes in Albumin to Globulin ratio | Week 0, 4, and 8
  Experimental outcome examining the ratio of Albumin to Globulin via fasted whole blood samples
Changes in Blood Urea Nitrogen to Creatinine ratio | Week 0, 4, and 8
  Experimental outcome examining the ratio of Blood Urea Nitrogen to Creatinine via fasted whole blood samples
Changes in estimated Glomerular Filtration Rate | Week 0, 4, and 8
  Experimental outcome examining the Glomerular Filtration rate via fasted whole blood samples
Changes in total mass | Week 0, 4, and 8
  Total mass will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Lean Body Mass | Week 0, 4, and 8
  Total lean body mass will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Fat Mass | Week 0, 4, and 8
  Total fat mass will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Bone Mineral Content | Week 0, 4, and 8
  Bone mineral content will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Bone Mineral Density | Week 0, 4, and 8
  Bone mineral density will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Body Fat Percentage | Week 0, 4, and 8
  Body Fat Percentage will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Body Mass Index | Week 0, 4, and 8
  Body Mass Index will be assessed via dual-energy x-ray absorptiometry (DEXA).
Changes in Grip Strength | Week 0, 4, and 8
  Assessed using a handheld dynamometer
Changes in Energy | Week 0, 4, and 8
  Assessed through a visual analog scale (100mm line), where 0 is no energy at all and 100 is very energized
Changes in Quality of Life | Week 0, 4, and 8
  Assessed by administering the Quality of Life Short Form (SF-36) for subjective measurement. Values range from 1 to 6 with higher scores demonstrating a better outcome.
Changes in Perceived Stress | Week 0, 4, and 8
  Assessed by administering the Perceived Stress Scale (PSS-10) for subjective measurement. Values range from 0 to 4 with lower scores demonstrating a better outcome.
Changes in Sleep Quality | Week 0, 4, and 8
  Assessed by administering the Sleep Quality Index (PSQI) for subjective measurement. Values range from 0 to 3 with lower scores demonstrating a better outcome.
Changes in Fatigue | Week 0, 4, and 8
  Assessed by administering the Multidimensional Fatigue Index for subjective measurement. Values range from 1 to 5 with lower scores demonstrating a better outcome.
Changes in Physical Activity | Week 0, 4, and 8
  Assessed by administering the International Physical Activity Questionnaire (IPAQ) for subjective measurement. Values are calculated by converting participant answers on time and intensity of physical activity to MET minutes with higher scores demonstrating a better outcome.

OTHER OUTCOMES:
Resting Systolic Blood Pressure | Week 0, 4, and 8
  Change in resting systolic blood pressure
Resting Diastolic Blood Pressure | Week 0, 4, and 8
  Change in resting diastolic blood pressure
Adverse Effects | Week 0, 4, and 8
  Defined as participants self-reported adverse effects. Items that will be surveyed are headache, dizziness, nausea, vomiting, indigestion, blurred vision, lethargy, swelling, itching, chest pain, heart palpitations, difficulty breathing, lethargy, and muscle cramps.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science and Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No